CLINICAL TRIAL: NCT02729857
Title: Postprandial Response After Intake of Meals With Different Fatty Acid Composition in Patients With Familial Hypercholesterolemia and Healthy Subjects
Brief Title: Postprandial Response After Intake of Meals With Different Fatty Acid Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Mills DA (Industry)
Responsible Party: Principal Investigator, Kirsten Holven, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015/2392/REK sør-øst B
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Healthy; Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Familial hypercholesterolemia (Experimental): Subjects diagnosed with familial hypercholesterolemia receive in randomized order muffin with saturated fat (SFA muffin) and polyunsaturated fat (PUFA muffin) at baseline
  Interventions: Dietary Supplement: SFA muffin; Dietary Supplement: PUFA muffin
- Healthy (Active Comparator): Subjects with no chronic diseases receive in randomized order muffin with saturated fat (SFA muffin) and polyunsaturated fat (PUFA muffin) at baseline
  Interventions: Dietary Supplement: SFA muffin; Dietary Supplement: PUFA muffin

INTERVENTIONS:
Dietary Supplement: SFA muffin — Muffin rich in saturated fat.
Dietary Supplement: PUFA muffin — Muffin rich in polyunsaturated fat.

SUMMARY:
The aim of the study is to understand more about how different fatty acids modulate postprandial lipid metabolism and inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 30 years of age
* Healthy or diagnosed with familial hypercholesterolemia (FH) (mutation in gene coding for LDL-receptor). FH subjects can be included if they are:

  1. Untreated
  2. Treated with low dose statin (<20 mg atorvastatin, <10-20 mg simvastatin or <5-10 mg rosuvastatin)
  3. Treated with high dose statin and willing to use low dose statin during the last 4 weeks prior to both study visits (total 8 week period)
  4. Treated with high dose statins and willing to discontinue statin treatment during the last 4 weeks prior to both study visits (total 8 week period)
* BMI 18.5 - 30 kg/m2
* Stabile weight the last three months prior to the first study visit (weight change less than ± 5 % of body weight)

Exclusion Criteria:

* CRP >10 mg/L
* TG >4 mmol/L
* Comorbidities including diabetes type I and II, coronary heart disease, haemophilia, anaemia, gastro intestinal disease, renal failure and hyperthyroidism
* Pregnant or lactating
* Allergic or intolerant to gluten or egg
* Not willing to stop using n-3 fatty acid supplements during the last 4 weeks prior to both study visits
* Using medications affecting lipid metabolism or inflammation, except statins for FH subjects
* Hormone treatment (except contraception and thyroxin (stabile dose last 3 months))
* Donating blood 2 months within or during study period
* Tobacco smoking
* Large alcohol consumption (>40g daily)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in levels of circulating triglycerides | Measured at baseline and 2,4 and 6 hours after intake of test meal

SECONDARY OUTCOMES:
Changes in markers of lipid- and glucose metabolism | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in levels of total cholesterol, low-density lipoprotein, high-density lipoprotein, apolipoprotein (apo) B, apo A1, apo CIII, apo B48, lipoprotein (a), free fatty acids, total fatty acid composition, LDL-receptor-related protein with 11 ligand-binding repeats (LR11), HbA1c, glucose, insulin and troponin.
Changes in circulating levels of inflammatory markers | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in levels of inflammatory markers in circulation such as i.e. cytokines and hsCRP
Changes in PBMC gene expression levels of markers of inflammation and lipid metabolism | Measured at baseline and 2, 4 and 6 hours after intake of test meal
  Changes in levels of markers of inflammation and lipid metabolism at PBMC gene expression level
Changes in lipid classes and lipoprotein size | Measured at baseline and 2,4 and 6 hours after intake of test meal
Changes in plasma and urine metabolomics | Measured in plasma at baseline and 2,4 and 6 hours after intake of test meal. Measured in urine at fasting state and during the 6 hour postprandial phase.
  Changes in metabolites such as glucose, lactate, pyruvate, citrate and amino acids will be measured in plasma and urine.
Check DNA for single nuclear polymorphisms | Measured at baseline and 2,4 and 6 hours after intake of test meal
Changes in PBMC Whole genome transcriptomics | Measured at baseline and 4 and 6 hours after intake of test meal

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Bjørklund Holven, Professor, Principal Investigator — Institute of Basic Medical Sciences, Faculty of medicine, University of Oslo
Locations (1):
- University of Oslo, Oslo, Post Box 1046, Blindern, Norway

IPD SHARING:
Plan to Share IPD: No